CLINICAL TRIAL: NCT05014152
Title: Prospective Trial for Clinical Validation of "QOCA Disposable BLE Thermometer "
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Quanta Computer Inc. (Unknown)
Responsible Party: Principal Investigator, Chih-Jung Chen, MD, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: QOCA-01
Record Dates: First submitted 2021-08-13; First posted 2021-08-20 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Fever
MeSH Terms: conditions — Fever

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (Experimental): This study is specially designed according to its age range and customized/non-customized range, and meets the requirements of ISO 80601-2-56 test population (table). Comply with the age range and population requirements of ISO 80601-2-56, as well as clinical and subject trials, including news to the population over five years old, and hopefuls must account for at least 30% of the total and less than 50% of the total.
  Each subject uses Q-temp-w1 to measure axillary temperature and obtains 3 temperature values, and at the same time uses a reference body temperature patch (Omron thermometer MC-171W) to measure the other side axillary temperature, and 1 is measured Temperature value data. Perform clinical efficacy analysis based on the measurement results. The main evaluation indicators of the trial include clinical bias, limits of agreement, and clinical repeatability.
  Interventions: Device: Q-temp-w1; Device: Omron thermometer(MC-171W)

INTERVENTIONS:
Device: Q-temp-w1 — Q-temp-w1 is a contact type body temperature patch developed by Quanta Computer Co., Ltd. It is mainly used to measure the body temperature of the human body. It can be used for general body temperature measurement, home temperature measurement records and medical tracking.
Device: Omron thermometer(MC-171W) — Omron thermometer(MC-171W) is mainly used to measure the body temperature of the human body. The reference temperature patch used in this study is the OMRON thermometer, model: MC-171W.

SUMMARY:
The purpose of this trial is to evaluate the accuracy and safety of the "QOCA Disposable Body Temperature Patch" (Q-temp-w1).

DETAILED DESCRIPTION:
Q-temp-w1 is a contact type body temperature patch developed by Quanta Computer Co., Ltd. It is mainly used to measure the body temperature of the human body. It can be used for general body temperature measurement, home temperature measurement records and medical tracking. Both the European Union and the US FDA state that the clinical test methods of the temperature patch must comply with ISO 80601-2-56. Therefore, this test plan will follow the ISO 80601-2-56 criteria to evaluate the accuracy of the temperature patch and follow it. The sampling age range and the fever/non-fever ratio are stratified, and clinical efficacy analysis is performed based on the measurement results. The main evaluation indicators include clinical bias, limits of agreement, and clinical repeatability.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female aged between 0-100 years.
* 2. Patient agrees to participate in the trial and sign informed consent.

Exclusion Criteria:

* 1. Those who have any broken skin or skin diseases on the part of the body which is the test site of the BLE thermometer, Including the underarms and the back of the body.
* 2. Those whose test site of the BLE thermometer are known to be contaminated by uncle arable body fluids, or lead to the inaccurate of the BLE thermometer.
* 3. Those who have restlessness or other conditions that make them unable to tolerate the temperature measurement procedure.

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Clinical bias | 10 min
  Use the first value of the 3 test patch body temperature data to calculate and analyze the paired data of the test subject with the reference body temperature data.

SECONDARY OUTCOMES:
Safety /Adverse Event Outcome Measure | 20 min / 24 hour (until recovered if it's SAE)
  Number of Participants with Serious and Non-Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Jung Chen, MD, Principal Investigator — Chang Gung Medical Fundation
Locations (1):
- ChangGungMH, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No